CLINICAL TRIAL: NCT03543488
Title: Neuromusuclar Responses and Functional Outcomes in Middle-aged Women With Rheumatoid Arthritis.
Brief Title: Neuromusuclar Adaptations in the Rheumatoid Arthritis Disease
Status: Completed | Type: Observational
Sponsor: Federal University of Rio Grande do Sul (Other)
Collaborators: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Principal Investigator, Marco Aurélio Vaz, PhD, Principal investigator, Federal University of Rio Grande do Sul
Other Study IDs: 09634
Record Dates: First submitted 2018-05-08; First posted 2018-06-01 (Actual); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Arthritis, Rheumatoid; Muscular Weakness
MeSH Terms: conditions — Arthritis, Rheumatoid; Muscle Weakness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Rheumatoid Arthritis Patients: Forty women (range 25-75 years), with a class I and II RA diagnosis according to the American Rheumatism Association's 1987 revised criteria, were recruited from a university hospital's rheumatology clinic. Exclusion criteria included the presence of any cardiovascular, neuromuscular and metabolic diseases or severe limitations in mobility. Five patients were excluded for not attending the inclusion criteria, leading to a final number of 35 RA patients.
  Interventions: Diagnostic Test: Neuromuscular and functional capacity tests
- Healthy Women: Thirty-five healthy women, age- and body size-matched to the RA patients, were recruited as controls (CG).
  Interventions: Diagnostic Test: Neuromuscular and functional capacity tests

INTERVENTIONS:
Diagnostic Test: Neuromuscular and functional capacity tests — The Timed Up and Go test; Maximal knee-extensor muscle strength (isometric and concentric tests) was measured with a Biodex System 3 dynamometer; A B-mode ultrasonography system with a linear-array probe (60 mm, 7.5 MHz) was used to determine VL and RF muscle thickness, pennation angle, fascicle length and tendon CSA. Measurements were obtained with the volunteer seated in the dynamometer, during isometric contraction at 90° of knee flexion.
  An 8-channel EMG system was synchronized with the dynamometer through a Windaq data acquisition system and used to evaluate the vastus lateralis and rectus femoris electrical activity during isometric knee-extensor tests.

SUMMARY:
Rheumatoid arthritis (RA) is a chronic autoimmune disease that causes joint inflammation and progressive joint destruction. Rheumatoid cachexia is one of the structural manifestations of RA, and consists of a reduction in muscle mass, due to an increased muscle protein catabolism induced by inflammatory cytokines. This muscle mass loss generates an impairment in physical function and functional capacity in RA patients. The aim of study was to verify neuromuscular and functional responses in middle-aged women with RA compared to paired healthy women.

ELIGIBILITY:
Inclusion Criteria:

* RA patients with a class I and II RA diagnosis according to the American Rheumatism Association's 1987 revised criteria, were recruited from a university hospital's rheumatology clinic.

Exclusion Criteria:

* presence of any cardiovascular, neuromuscular and metabolic diseases or severe limitations in mobility

Ages: 25 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 35 RA patients (class I and II according American Rheumatism Association) and 35 healthy women, age- and body size-matched to the RA patients, were recruited as controls (CG).
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2013-06-01 (Actual); Primary Completion 2013-11-20 (Actual); Study Completion 2014-03-03 (Actual)

PRIMARY OUTCOMES:
Knee-Extensor Muscular Strength | Only one day.
  Maximal knee-extensor muscle strength (isometric and concentric tests), in different angles and velocities were measured with a Biodex System 3 dynamometer (Biodex Medical Systems, Shirley, NY, USA). A 2-min interval was observed between contractions. We used the peak torque of each maximal test to analysis.
Muscle architecture and tendon parameters | Only one day.
  An ultrasonography system was used to determine VL and RF muscle thickness, pennation angle and fascicle length. Muscle architecture measurements were obtained with the volunteer seated in the dynamometer, during isometric contraction at 90° of knee flexion. Muscle thickness was considered the distance between deep and superficial aponeuroses. The best fascicle in each image was used for pennation angle and fascicle length analysis. Pennation angle was calculated as the angle between the muscle fascicle and the deep aponeurosis, whereas fascicle length was measured as the length of the fascicular path between the two aponeuroses. Furthermore, patellar tendon cross-section area was measured with probe perpendicular to tendon during isometric contractions.
Functional Capacity | Only one day.
  Timed Up and Go test
Quadriceps muscle activation | Only one day.
  Vastus Lateralis and Rectus Femoris muscle activation during strength tests

IPD SHARING:
Plan to Share IPD: No